CLINICAL TRIAL: NCT05540873
Title: A Single-center, Single-arm, Open-label Phase 1 Clinical Trial to Assess the Safety and Tolerability of YYB-103, IL13Rα2 Targeted Chimeric Antigen Receptor-T Cell (CAR-T) in Treating Patients With Refractory or Recurrent Malignant Glioma
Brief Title: A Clinical Study of IL13Rα2 Targeted CAR-T in Patients With Malignant Glioma (MAGIC-I)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CellabMED (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLM_103_MG001
Record Dates: First submitted 2022-08-28; First posted 2022-09-15 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-09

CONDITIONS: Recurrent Malignant Glioma
Keywords: Chimeric antigen receptor; Malignant glioma; IL13Rα2; CLM_103_MG001; YYB103; MAGIC-I
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IL13Rα2 targeted CAR-T (Experimental)
  Interventions: Drug: YYB-103

INTERVENTIONS:
Drug: YYB-103 — Biological: IL13Rα2 CAR-T cells Administration method: intravenous infusion YYB-103 is manufactured according to the subject's assigned dose group and body weight.

SUMMARY:
This is a phase I study to evaluate the safety and tolerability of IL13Rα2 Targeted Chimeric Antigen Receptor-T Cell in patients with Refractory or Recurrent Malignant Glioma and to evaluate the changes of AE incidence.

And this study have to long term follow-up.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label phase 1 study that will follow a 3 + 3 design of dose-escalating cohorts. The objectives of this study is to assess the safety and tolerability after administration of YYB-103 (IL13Rα2 targeted CAR-T cell) in patients with malignant glioma.

YYB-103 is designed to target cancer cells expressing IL13Rα2 in cell surface. Only those subjects who are expressing IL13Rα2 and satisfy the inclusion and exclusion criteria will receive IV infusion of YYB-103.

Long term follow-up study is evaluate the safety and exploratory efficacy of IP for 15 years from the date of IP administration in patients with malignant glioma refractory or recurrent to standard therapy who participated in this study.

Subjects who participated in the Phase 1 study and received YYB-103 must have long-term follow-up for 15 years from the date of administration. During the long-term follow-up period, AEs, exploratory efficacy etc. are observed, and the observation period is every 6 months within 5 years and then yearly until 15 years.

ELIGIBILITY:
Inclusion Criteria

1. Primary inclusion criteria (Screening criteria)

   : Only subjects who meet all of the following conditions conduct examinations and tests including the IHC and PBMC
   * Provision of voluntary written consent to participate in this clinical trial
   * Male and female aged ≥ 19 years to <75 years
   * Patients with histologically or cytologically confirmed progressive malignant glioma (Grade III or IV according to the WHO criteria) and histological and/or radiologic data to confirm that it is refractory or recurrent (applicable to 'Progression Disease (PD)' according to the Response Assessment for Neuro-Oncology (RANO) criteria for high grade gliomas defined by the Society for Neuro-Oncology) despite treatment applicable to the standard treatment for each stage
   * Subject with the Karnofsky Performance Status (KPS) Scale ≥ 60
   * Subject with the life expectancy of least 12 weeks at the investigator's discretion
   * Subject who satisfies the following treatment condition, regardless of the previous line of treatment
   * At least 12 weeks after completion of the last anticancer radiation treatment
   * Other cell toxicity therapy not mentioned above: At least 3 weeks have passed
   * Non-cytotoxic agent (e.g., interferon, tamoxifen, etc.): At least 1 week has passed
   * Completion of treatment of all toxicities and AEs (other than alopecia and vitiligo) due to the previous treatment
2. Secondary Inclusion Criteria (Eligibility Criteria)

   * Subjects confirmed as positive for IL13Rα2 expression from immunostaining (IHC)
   * Subjects with Peripheral Blood Monocyte Count ≥ 7.5x10^5 cells/5 ml from the PBMC test
   * Subjects with appropriate bone marrow, liver, and kidney function by satisfying all of the following in clinical laboratory tests

     * WBC ≥ 2,000/μl
     * ANC ≥ 1,000/μl
     * Platelet count ≥ 75,000/μl
     * Hemoglobin ≥ 8.0 g/dL
     * ALT/AST ≤ 2.5 x ULN
     * Serum creatinine ≤ 1.5 x ULN
     * Total bilirubin ≤ 1.5 x ULN

Exclusion Criteria

1. Primary Exclusion Criteria (Screening criteria)

   * Subjects diagnosed with ventricular seeding, spinal drop metastasis, or leptomeningeal metastasis from radiologic testing obtained at screening
   * Subjects with findings of immunodeficiency, autoimmune disease (e.g.; rheumatoid arthritis, systemic lupus erythematosus, vasculitis, multiple sclerosis, etc.) or inflammatory disease
   * Subjects with significant active cardiovascular disease including the following

     * Uncontrolled hypertension (SBP >180 mmHg or DBP >110 mmHg), unstable angina, pulmonary embolism, cerebrovascular disease, valvular disease, cardiac failure, or myocardial infarction or serious cardiac arrhythmia within the past 6 months
   * Subjects with a medical history of malignant tumor other than the study indication within 5 years of screening (however, within 3 years of screening in case of malignant tumor (e.g., appropriately treated cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ, etc.) with minimal risk of metastasis/recurrence and death)
   * Subjects who continuously used systemic immunosuppressants (including but not limited to cyclophosphamide, azathioprine, methotrexate, and thalidomide) other than steroids within 2 weeks of screening
   * Subjects on systemic steroids who received a dose exceeding dexamethasone 6 mg/day (or equivalent dose) within 1 week of screening(note that topical steroids, inhaled steroid, and use of transient steroids for prevention of vomiting prior to anticancer agents administration are acceptable)
   * Subjects with a history of previously using an immune cell therapy agent
   * Subjects with a medical history of severe allergy, anaphylaxis, or other hypersensitivity reaction to the chimeric or humanized antibody or fusion protein
   * Subjects who participated in other clinical trial (medicinal product or medical device) within 4 weeks of screening
   * Women of childbearing potential and men who have a plan to get pregnant until 3 months after investigational product administration, are not willing to practice appropriate contraception method*, or are not willing to maintain abstinence from sexual intercourse

     * Hormonal contraception method, intrauterine device (IUD) or intrauterine system (IUS), surgical sterilization of the subject or partner, tubal ligation, double barrier method (a combined use of a barrier method such as a female condom, cervical cap, contraceptive diaphragm, or contraceptive sponge with a male condom), single barrier method combined with spermicide)
   * Pregnant women or breastfeeding mothers
   * Subjects who are determined by the investigator to be ineligible as subjects of this clinical trial for other reason
2. Secondary Exclusion Criteria (Eligibility Criteria)

   * Subjects who are positive to any of the following virus test results at screening

     * Hepatitis B virus surface antigen (HBsAg)
     * Hepatitis C virus antibody test (anti-HCV Ab)
     * HIV antibody test (anti-HIV)
   * Subjects who are determined by the investigator to be ineligible as subjects of this clinical trial for other reason

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 28 days after IP administration
Maximum Tolerance Dose (MTD) | 28 days after IP administration
Recommended Phase 2 Dose (RP2D) | 28 days after IP administration

SECONDARY OUTCOMES:
Incidence of AE | 3 months, up to 15 years if necessary
  CRS and ICANS (ASTCT) / Others (CTCAE V5.0)
RCR | 1 year, up to 15 years if necessary
  RCR formation will be checked by collecting samples at 3M, 6M, and every 6 months thereafter until 5 years from IP administration, and then will be followed up annually thereafter until 15 years from IP administration via medical history without collecting samples. If all RCR test results are negative for 1 year after IP administration, sample collection will be stopped, and annual follow-up.
Pharmacokinetics and cytokine levels | 3 months, up to 15 years if necessary
  Peripheral blood (PB) and Cerebral spinal fluid (CSF)
Disease response (DCR) | Baseline up to 6 months
  Tumor response will be assessed by comparison with baseline magnetic resonance imaging by iRANO criteria. Evaluation of DCR is the proportion of subjects with CR or PR or SD as a result of tumor response assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea